CLINICAL TRIAL: NCT07224295
Title: The Effect of Non Invasive Stellate Ganglion Disrupting on Sleep Disturbances on Postmenopausal Female
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Wafaa Shaaban Hassan Elbeltagy, Senior physical therapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-765
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Sleep Disturbances
MeSH Terms: conditions — Parasomnias | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: TENS (Frequency 80 _100 Hz), (Pulse duration: 150-200 μs, Pain-free stimulation intensity), (Duration;30 min)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): TENS Application
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Dietary Supplement: Lactium
- Group 2 (Experimental): Lactium
  Interventions: Dietary Supplement: Lactium

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS (Frequency 80 _100 Hz), (Pulse duration: 150-200 μs, Pain-free stimulation intensity), (Duration;30 min) On one side of the patient's neck, at the location of the stellate ganglion, we positioned two adhesive 25 mm to administer the TENS treatment, while the other side remained untreated. Of the two adhesive electrodes, one was placed near to the paravertebral location in the region of the trapezius muscle on its base near the sixth cervical transverse process, and the other in the region of the stellate ganglion in the supraclavicular aspect (Fig. 2). To obtain a stellate ganglion disrupting, we used a dual-channel TENS stimulator.
  Arms: Group 1
Dietary Supplement: Lactium — Lactium is a natural milk protein hydrolysate that contains a bioactive decapeptide called alpha-casozepine, which has natural relaxing and calming properties. It is used as a dietary supplement ingredient to help manage symptoms of stress, anxiety, and sleep disorders.this supplement will be taken once daily

SUMMARY:
The goal of this clinical trial is to asses the effect of non invasive stellate ganglion disrupting on sleep distyrbances on postmenopausal female .

The primary hypothesis:

There is no effect of noninvasive stellate ganglion disrupting on sleep disturbance parameters of postmenopausal women.

There is no effect of noninvasive stellate ganglion disrupting on quality of female's life

Non invasive stellate ganglion disrupting with physical modality TENS will be applied on participants of study group. The participants will be screened for estradiol level and assed for the quality of sleep by specialized questionnaire.

DETAILED DESCRIPTION:
This study will be conducted on 32 postmenopausal women referred by physicians having sleep disturbances. They will be recruited from kafr el-zayat General Hospital, El-gharbia Governorate, Egypt.

All participants will be given a full explanation of the protocol of the study and informed consent form will be signed from each subject before participating in this study. The protocol will be sent for approval the ethical committee of the faculty of Physical Therapy kafrelshekh University.

The subjects will be divided randomly into two groups equal in number, study group (group A) and control group (group B):

* Study group (group A): This group will consist of sixteen women complaining from sleep disturbance with post menopause who will receive TENS (Frequency 80 _100 Hz), (Pulse duration: 150-200 μs, Pain-free stimulation intensity), (Duration;30 min).
* Control group (group B): This group will consist of sixteen women complaining from sleep disturbance with post menopause.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal women who are firstly have sleep disturbances.
2. Their ages will range from 50- 65 years old.
3. All patients will be medically stable when attending the study.
4. BMI≥30.

Exclusion Criteria:

-

Women will be excluded from study if:

1. Women with Impaired consciousness.
2. Inability to communicate with the paramedic because of insufficient language skills.
3. receiving any medication for sleep disturbances.
4. Patients who already have sleep disturbances due to another pathological reason or taking any medications which directly affect sleep.
5. Patients with psychological diseases.
6. Women who have any cancer diseases.
7. Diabetic and patient with cardiovascular disease.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post menopausal female
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of estradiole plasma level | After 3 months of treatment
  by biochemical examination of estradiole plasma level
Change of sleep quality | After 3 months of treatment
  By assesment of the global pittsburgh sleep quality index scores a self-rated sleep questionnaire, were used to measure the quality of sleep. There are seven different parts that add up to a total of 19 questions. The scores range from 0 (no difficulty) to 3 (severe difficulty). The components include subjective sleep quality, sleep latency, length, and normal efficiency of sleep; they also include sleep disruptions, use of sleep medications, and dysfunction during the day. The seven component scores are also added together to create a global Pittsburgh Sleep Quality Index score, which ranges from 0 to 21. A score of more than 5 indicates a clinical sleep disability.

CONTACTS AND LOCATIONS:
Overall Officials: fayez f Elshamy, professor, Principal Investigator — kafrelshekh university
Locations (1):
- Wafaa shaaban hassan elbeltagy, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No